CLINICAL TRIAL: NCT05018494
Title: Effects Of Supervised Sensorimotor Training With And Without Lifestyle Modifications Through Telerehabilitation Monitoring After Total Knee Arthroplasty
Brief Title: Effects Of Supervised Sensorimotor Training Through Telerehabilitation Monitoring After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/2033
Record Dates: First submitted 2021-08-12; First posted 2021-08-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Arthropathy of Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group will receive the common treatment and will be discharged with complete manual on life style modifications comprising education, exercise and diet with telerehabilitation monitoring.
  Interventions: Other: experimental treatment
- Group B (Active Comparator): This group will receive the common treatment and will be discharged with home exercise plan without telerehabilitation monitoring.
  Interventions: Other: common treatment

INTERVENTIONS:
Other: experimental treatment — This group will receive the common treatment and will be discharged with complete manual on life style modifications comprising education, exercise and diet with telerehabilitation monitoring.
  Arms: Group A
Other: common treatment — This group will receive the common treatment and will be discharged with home exercise plan without telerehabilitation monitoring.
  Arms: Group B

SUMMARY:
Knee Osteoarthritis (OA) along with low back pain, is one of the most frequent rheumatic disorder in the Asian regions. Total Knee Arthroplasty is considered as a gold standard management strategy for relieving symptoms due to degenerative arthritis of knee. Rehabilitation after knee arthroplasty is an essential component among this population and plays a significant role in improving the functional performance and quality of life. However, access to rehabilitation, health care services and follow up is not always possible. One of the possible solution is the utilization of telerehabilitation technology to allow monitoring facilities be delivered to the patients from distance, so that follow up of a patient could be ensured. Secondly, a type of therapeutic exercise followed after knee replacement constitutes muscle strengthening, muscle stimulation with resistance exercises, sensorimotor training and telerehabilitation. Sensorimotor training improves central nervous system function for managing movement and appropriate muscular firing patterns for maintaining joint stability. An important component missing in the treatment regime of a knee replacement patient is the lifestyle modification program which is a combination of education, exercise and diet. So, the aim of current project is to evaluate the effects of supervised sensorimotor training with and without lifestyle modifications through telerehabilitation monitoring on joint position sense, balance, posture, muscle strength, knee joint function and quality of life after total knee arthroplasty. The telerehabilitation system would interaction between clinician at hospital and patients at home. A web based portal will be developed and then utilized to provide the user with personalized information such as guided video and audio instructions about each exercise. The digital rehabilitation solution is well established in developed nations. It is the need of hour to introduce technological advancements in Pakistan. Tele-rehabilitation should be incorporated as it will be helpful for the community and will reduce the dependence on human resources while ensuring better clinical outcomes as standard therapy. Intervention group will receive lifestyle modification manual and follow up will be ensured through telerehabilitation monitoring. Analysis will be done through SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female
2. Successful Total Knee Arthroplasty surgery
3. Ability to walk (with walking aid or unaided)
4. Aged between 45 to 75 years old,
5. Active knee flexion of 80 degree and active knee extension of -10 degree upon discharge
6. Availability of internet service in the residing area.

Exclusion Criteria:

1. Presence of health related medical conditions that could interfere with tests or the rehabilitation program
2. Neurological conditions that might affect balance
3. Inability to attend rehabilitation services, revised knee arthroplasty
4. Blindness and any condition incompatible with 30 minutes of light to moderate physical activity

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Joint position sense | 6 months
  through digital photography and timings will be measured the difference between the 3 repetition will be measured. error will be measured in seconds through photographic software.
Muscle thickness of Rectus femoris | 6 months
  through ultrasound. as muscle relax it will lengthen it will measured in mili meters
Berg balance scale | 6 months
  The berg balance scale (BBS) consists of 14 items scored on a 5-point ordinal scale, ranging from 0 to 4 (0 indicates lowest level of function; 4 indicates highest level of function), with a maximum total score of 56. Participants presenting a score of 41 to 56 points have been described as "independent"; scores of 21 to 40 are interpreted as "walking with assistance"; and scores of 0 to 20 are generally classified as "wheelchair bound."
knee function | 6 months
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a self-administered health status measure that assesses the dimensions of pain, stiffness and function The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.
Quality of life (SF 12) | 6 months
  SF 12 Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning [27]. A score of 50 or less on the PCS-12 has been recommended as a cut-off to determine a physical condition; while a score of 42 or less on the MCS-12 may be indicative of 'clinical depression

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Lahore Medical and Dental College, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iqbal MN, Haidri FR, Motiani B, Mannan A. Frequency of factors associated with knee osteoarthritis. J Pak Med Assoc. 2011 Aug;61(8):786-9. PMID 22356003
- [Background] Kuether J, Moore A, Kahan J, Martucci J, Messina T, Perreault R, Sembler R, Tarutis J, Zazulak B, Rubin LE, O'Connor MI. Telerehabilitation for Total Hip and Knee Arthroplasty Patients: A Pilot Series with High Patient Satisfaction. HSS J. 2019 Oct;15(3):221-225. doi: 10.1007/s11420-019-09715-w. Epub 2019 Aug 21. PMID 31624476
- [Background] Tousignant M, Moffet H, Boissy P, Corriveau H, Cabana F, Marquis F. A randomized controlled trial of home telerehabilitation for post-knee arthroplasty. J Telemed Telecare. 2011;17(4):195-8. doi: 10.1258/jtt.2010.100602. Epub 2011 Mar 11. PMID 21398389
- [Background] Wadden TA, Butryn ML, Wilson C. Lifestyle modification for the management of obesity. Gastroenterology. 2007 May;132(6):2226-38. doi: 10.1053/j.gastro.2007.03.051. PMID 17498514
- [Background] Dalle Grave R, Calugi S, Centis E, Marzocchi R, El Ghoch M, Marchesini G. Lifestyle modification in the management of the metabolic syndrome: achievements and challenges. Diabetes Metab Syndr Obes. 2010 Nov 2;3:373-85. doi: 10.2147/DMSOTT.S13860. PMID 21437107